CLINICAL TRIAL: NCT04314765
Title: Clinical Wound Healing After Fully-impacted Lower Third Molar Surgery Using Two Different Type of Flap: Randomized Clinical Trial
Brief Title: Clinical Wound Healing After Lower 3rd Molar Fully-impacted Surgery With 2 Types of Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Pippi Roberto, MDDS, associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5478/25.7.19
Record Dates: First submitted 2020-03-10; First posted 2020-03-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-04

CONDITIONS: Wound Heal; Quality of Life; Dehiscence
Keywords: third molar surgery; flaps; health related quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bayonet flap (Experimental): Bayonet flap is performed to extract the the lower third molar
  Interventions: Procedure: lower third molar extraction
- envelope flap (Experimental): Envelope flap is performed to extract the the lower third molar
  Interventions: Procedure: lower third molar extraction

INTERVENTIONS:
Procedure: lower third molar extraction — the extraction is performed with one of the two type of flap based non randomization.

SUMMARY:
The dehiscence distal to the second molar after lower third molar extraction is very common because the access flap for surgical extraction cannot be repositioned on a portion of healthy bone to guarantee suture support. The healing process is therefore delayed and the possible accumulation of food and debris is often responsible for bad smell and pain with the consequent occurrence of an overlapping infection.

The main aim of the study is to evaluate whether healing is significantly different using two different flaps for surgical access. Clinical assessment and a quality of life questionnaire are used for the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* fully-impacted lower third molar
* patients aged between 18 and 35

Exclusion Criteria:

* patients undergoing drug treatment for systemic diseases that can influenced the healing process,
* pregnant women,
* smoking habits
* patients with disabilities
* all interventions in which intraoperative accidents involving the soft tissues occurred (laceration of the mucosa / flap).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
wound healing day 2 | 2 days after surgery
  a clinical chart is complete to evaluate if in the group of lower third molar extracted with a bayonet flap the proportion of healing without dehiscence (good healing index) is significant greater than in the group of third molar extracted with an envelope flap.
wound healing day 7 | 7 days after surgery, at suture removal
  a clinical chart is complete to evaluate if in the group of lower third molar extracted with a bayonet flap the proportion of healing without dehiscence (good healing index) is significant greater than in the group of third molar extracted with an envelope flap.
wound healing day 14 | 14 days after surgery
  a clinical chart is complete to evaluate if in the group of lower third molar extracted with a bayonet flap the proportion of healing without dehiscence (good healing index) is significant greater than in the group of third molar extracted with an envelope flap.

SECONDARY OUTCOMES:
quality of life day 2 | 2 days after surgery
  the patient complete a HRQOL questionnaire (modify from Shugars DA et al 1996) to evaluate if differences exist in the patient's quality of post-operative life in relation with two types of flap; we use visual analog scales (VAS) for post-operative pain and five-points Likert-Type for swelling, chewing, speaking, sleeping, sport and daily routine activity; higher scores mean a worse outcome.
quality of life day 5 | 5 days after surgery
  the patient complete a HRQOL questionnaire (modify from Shugars DA et al 1996) to evaluate if differences exist in the patient's quality of post-operative life in relation with two types of flap; we use visual analog scales (VAS) for post-operative pain and five-points Likert-Type for swelling, chewing, speaking, sleeping, sport and daily routine activity; higher scores mean a worse outcome.
quality of life day 7 | 7 days after surgery, at suture removal
  the patient complete a HRQOL questionnaire (modify from Shugars DA et al 1996) to evaluate if differences exist in the patient's quality of post-operative life in relation with two types of flap; we use visual analog scales (VAS) for post-operative pain and five-points Likert-Type for swelling, chewing, speaking, sleeping, sport and daily routine activity; higher scores mean a worse outcome.
quality of life day 14 | 14 days after surgery
  the patient complete a HRQOL questionnaire (modify from Shugars DA et al 1996) to evaluate if differences exist in the patient's quality of post-operative life in relation with two types of flap; we use visual analog scales (VAS) for post-operative pain and five-points Likert-Type for swelling, chewing, speaking, sleeping, sport and daily routine activity; higher scores mean a worse outcome.
dehiscence | 2 days after surgery
  a clinical chart is complete to evaluate if the presence of the dehiscence makes differences in surgical wound healing
dehiscence | 7 days after surgery, at suture removal
  a clinical chart is complete to evaluate if the presence of the dehiscence makes differences in surgical wound healing
dehiscence | 14 days after extraction
  a clinical chart is complete to evaluate if the presence of the dehiscence makes differences in surgical wound healing
pre-operative symptoms | pre-operative
  the presence or not of pre operative Symptoms
interincisive height | pre-operative
  the distance between upper and lower central incisors
Full Mouth Plaque Score | pre-operative
  Full-mouth plaque score was recorded dichotomously (presence/absence of plaque) on six sites per tooth and was then calculated as the percentage of total tooth surfaces that revealed the presence of plaque; higher percentage mean higher presence of plaque
Partial Plaque Score | pre-operative
  Partial plaque score was recorded dichotomously (presence/absence of plaque) on six sites per tooth in the arch of extraction and was then calculated as the percentage of total tooth surfaces that revealed the presence of plaque; an higher percentage means higher presence of plaque
type of impaction | pre-operative
  on orthopantomography
Pell & Gregory class | intra-operative
  on orthopantomography
depth of impaction | pre-operative
  on orthopantomography
tooth position | pre-operative
  on orthopantomography
description root morphology | pre-operative
  on orthopantomography; apical anomalies yes/no
description number of roots | pre-operative
  on orthopantomography; 1/2/3/more than 3
description of relationship with the second molar | pre-operative
  on orthopantomography; no contact/contiguity/overlap
probing depth distal to the second molar | pre-operative
quantity of keratinized gingiva | pre-operative
position of the gingiva with respect to the CEJ (cemento-enamel junction) of the second molar | pre-operative
maximum diameter of the bone cavity | intra-operative
maximum depth of the bone cavity | intra-operative
  maximum depth of the bone cavity with respect to the CEJ of the second molar
position of the gingiva | intra-operative
  position of the gingiva after the suture with respect to the CEJ (cemento-enamel junction) of the second molar
duration of surgery | intra-operative
  extraction and suture

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pippi, MDDS, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Pippi Roberto, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No